CLINICAL TRIAL: NCT00308360
Title: Risperidone Alone Vs. Risperidone Plus Valproate in the Treatment of Patients With Schizophrenia and Hostility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Janssen, LP (Industry); Research Foundation for Mental Hygiene, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIS-189; RIS-189
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2006-03-29 (Estimated); Status verified 2006-03

CONDITIONS: Schizophrenia
Keywords: Hostility; Impulsivity; Aggression
MeSH Terms: conditions — Schizophrenia; Impulsive Behavior; Aggression | interventions — Risperidone; Valproic Acid

INTERVENTIONS:
Drug: Risperidone, divalproex

SUMMARY:
This is an eight-week open-label randomized parallel group clinical trial focusing on the comparison of risperidone alone with risperidone plus valproate among hospitalized adult patients diagnosed with schizophrenia who also exhibit problems with hostility. Patients may have already been receiving risperidone or valproate (but not both) at study entry. Patients not receiving valproate at study entry were randomized to receive either risperidone alone or risperidone with valproate. For patients already receiving valproate at study entry, their antipsychotic medication(s) was switched to risperidone, and they were followed for a four-week lead-in period prior to baseline assessment and randomization to receive risperidone alone or continue with risperidone and valproate. We hypothesized that risperidone alone has an antiaggressive/antihostility effect, and that this effect is augmented by the co-administration of valproate.

DETAILED DESCRIPTION:
Background: Patients with schizophrenia who also exhibit hostile behavior pose a formidable challenge for clinicians. Hostile behavior is a frequent reason for psychiatric admission, and is an obstacle for the successful reintegration of patients back into the community. Current treatment approaches have generally not been assessed under controlled conditions.

Method: This is an eight-week open-label randomized parallel group clinical trial focusing on the comparison of risperidone alone with risperidone plus valproate among hospitalized adult patients diagnosed with schizophrenia who also exhibit problems with hostility. Patients may have already been receiving risperidone or valproate (but not both) at study entry. Patients not receiving valproate at study entry were randomized to receive either risperidone alone or risperidone with valproate. For patients already receiving valproate at study entry, their antipsychotic medication(s) was switched to risperidone, and they were followed for a four-week lead-in period prior to baseline assessment and randomization to receive risperidone alone or continue with risperidone and valproate. Blinded raters completed a battery of assessments, including the Positive and Negative Syndrome Scale, Buss-Durkee Hostility Inventory, Barratt Impulsiveness Scale, and the Overt Aggression Scale. We hypothesized that risperidone alone has an antiaggressive/antihostility effect, and that this effect is augmented by the co-administration of valproate.

ELIGIBILITY:
Inclusion Criteria:

1) Male or female, age 18 to 65 inclusive, diagnosed with schizophrenia (not including schizoaffective disorder) according to DSM-IV criteria using the Structured Clinical Interview for DSM-IV Axis I Disorders; 2) Referral from the treating psychiatrist/treatment team because of difficulties with poor impulse control; 3) At study entry the subject must have scored at least "3" ("mild" or above) on at least one of the following Positive and Negative Syndrome Scale items that comprise the activation factor: Hostility, Impulsivity, Excitement, or Uncooperativeness; 4) Capacity and willingness to give informed consent; 5) Adequate knowledge of English; 6) Absence of serious medical illness; and 7) Accessible, adequate veins likely to permit repeated venipunctures without major problems.

Exclusion Criteria:

1) Receiving both adequate amounts of valproate and risperidone at the time the inclusion criteria have been met. This was defined as a dose of valproate that was equal to or exceeding 1000 mg/day (or a plasma level equal to or greater than 50 micrograms/mL) for at least 2 weeks, and any dose of risperidone; 2) History of severe adverse reaction to either risperidone or valproate; 3) Administration of a slow-release antipsychotic (depot) within 30 days preceding randomization; and 4) Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 1999-09; Study Completion 2004-04

PRIMARY OUTCOMES:
Buss-Durkee Hostility Inventory
Barratt Impulsiveness Scale

SECONDARY OUTCOMES:
Overt Aggression Scale
Positive and Negative Syndrome Scale

CONTACTS AND LOCATIONS:
Overall Officials: Leslie L Citrome, MD, MPH, Principal Investigator — Nathan S Kline Institute for Psychiatric Research and New York University School of Medicine; Jan Volavka, MD, PhD, Principal Investigator — Nathan S Kline Institute for Psychiatric Research and New York University School of Medicine
Locations (1):
- Nathan S Kline Institute for Psychiatric Research and Rockland Psychiatric Center, Clinical Research and Evaluation Facility, Orangeburg, New York, United States

REFERENCES:
- [Derived] Citrome L, Shope CB, Nolan KA, Czobor P, Volavka J. Risperidone alone versus risperidone plus valproate in the treatment of patients with schizophrenia and hostility. Int Clin Psychopharmacol. 2007 Nov;22(6):356-62. doi: 10.1097/YIC.0b013e3281c61baf. PMID 17917554
- See also: Nathan S Kline Institute for Psychiatric Research — http://www.rfmh.org/nki